CLINICAL TRIAL: NCT03135288
Title: Effect of Cell-phone Assisted Postpartum Counseling on the Use of Long-acting Reversible Contraceptives: a Randomized Controlled Trial
Brief Title: Cell-phone Assisted Postpartum Counseling on the Use of Long-acting Reversible Contraceptives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CP-LARC
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Family Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell-phone assisted (Experimental): will be advised that they are going to receive a reminder of their postpartum family planning visit 5 weeks after the delivery (one week before the scheduled visit) and a phone call 48 hours before the scheduled visit. They will also receive two follow-up phone calls to answer any questions and to remind them with the follow-up visits after insertion. Woman will be given a referral card to the outpatients' family planning clinic denoting her study group and serial number and with a specific date for postpartum family planning visits. They will be also provided with a cell phone number working 7 days a week to answer any query or questions regarding her family planning program.
  Interventions: Device: Cell-phone
- control group (No Intervention): will receive the same above adequate counseling with referral card but without any phone assistance

INTERVENTIONS:
Device: Cell-phone — a reminder of their postpartum family planning visit 5 weeks after the delivery (one week before the scheduled visit) and a phone call 48 hours before the scheduled visit. They will also receive two follow-up phone calls to answer any questions and to remind them with the follow-up visits after insertion. Woman will be given a referral card to the outpatients' family planning clinic denoting her study group and serial number and with a specific date for postpartum family planning visits.
  Arms: Cell-phone assisted

SUMMARY:
Unintended and closely spaced pregnancies are a major public health problem that affects not only the individuals directly involved but also the society indirectly. It increases the risks of infants with adverse outcomes such as preterm, low birth weight and small for gestational age. Pregnancy occurring within six months of the last delivery holds a 7.5-fold increased risk for induced abortion, a 3.3-fold increase in miscarriage and a 1.6-fold increased risk of stillbirth. But, use of contraceptive methods has been shown to reduce unwanted pregnancy, high fertility and maternal mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver a live birth at greater than 28 week's gestation.
* Women desire birth spacing for more than one year
* Women who were holding and /or one of her family hold a cell-phone and accept to receive messages and phone calls to remind her with her contraceptive program

Exclusion Criteria:

* Women who refuse to participate in the study.
* Women aren't able to respond to the questionnaire due to their health status.
* Anticipation of difficulty of subsequent communication with the women
* Women with contraindications of using long acting reversible contraception ( contraindicated if intrauterine device or implant use)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Initiation of Long acting reversible contraception method | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Shaaban OM, Saber T, Youness E, Farouk M, Abbas AM. Effect of a mobile phone-assisted postpartum family planning service on the use of long-acting reversible contraception: a randomised controlled trial. Eur J Contracept Reprod Health Care. 2020 Aug;25(4):264-268. doi: 10.1080/13625187.2020.1764528. Epub 2020 May 21. PMID 32436800